CLINICAL TRIAL: NCT00615394
Title: Autologous Transplantation of Bone Marrow Mononuclear Stem-Cells by Mini-Thoracotomy in Dilated Cardiomyopathy - Technique and Early Results
Brief Title: Autologous Transplantation of Bone Marrow Mononuclear Stem-Cells by Mini-Thoracotomy
Acronym: STEMDILCARD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Instituto de Cardiologia do Rio Grande do Sul / Fundação Universitária de Cardiologia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UP3549/04
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2008-02-14 (Estimated); Status verified 2008-02

CONDITIONS: Dilated Cardiomyopathy
Keywords: cardiomyopathy, stem cell, cardiac failure
MeSH Terms: conditions — Cardiomyopathy, Dilated; Cardiomyopathies; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: intramyocardial bone marrow stem cells implantation — Patients with previous diagnosis of non-ischemic dilated cardiomyopathy. were included. Bone-marrow was collected from in the antero-superior iliac crest and mononuclear stem-cells were isolated by centrifugation in the density rate Ficoll-Hypaque 1.077 media. Surgical technique - The approach was through a left mini-thoracotomy. Twenty small injections of cellular suspension were directly made through a 21F butterfly needle(total=5 ml), in the anterior, lateral, posterior and apical faces of the left ventricle(average 9.6 ± 2.6 x 107 cells). After the procedure, the patients were kept in the post-operative intensive care unit for a minimum period of 24 hours. They were released from the hospital in a period that varied from five to seven days.

SUMMARY:
Bone marrow mononuclear cells (BMMC) transplantation is a promising therapy for treating ischemic disease, however the effect in non-ischemic dilated cardiomyopathy is unknown.This study describes a technique of BMMC transplantation utilizing mini-thoracotomy and results up to one year after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis made at more than two years and symptomatic at functional class III-IV by the New York Heart Association classification (NYHA) despite optimal pharmacologic therapy
* left ventricular ejection fraction (LVEF) less than 35%, by echocardiogram
* age below 60 years
* absence of neoplasm
* absence of hematologic disease or systemic disease
* no previous cardiac intervention

Exclusion Criteria:

* episodes of tachycardia or ventricular fibrillation
* severe or moderated mitral insufficiency
* any other valvulopathies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2004-04; Primary Completion 2006-10 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
safety: morbidity/mortality | eighteen months

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Kalil RA, Ott D, Sant'Anna R, Dias E, Marques-Pereira JP, Delgado-Canedo A, Nardi NB, Sant'Anna JR, Prates PR, Nesralla I. Autologous transplantation of bone marrow mononuclear stem cells by mini-thoracotomy in dilated cardiomyopathy: technique and early results. Sao Paulo Med J. 2008 Mar 6;126(2):75-81. doi: 10.1590/s1516-31802008000200003. PMID 18553028